CLINICAL TRIAL: NCT02211898
Title: Clinical Study of BNS003 on Swelling Due to Disorder of Leg Venous Reflux
Brief Title: Clinical Study of BNS003 on Swelling in Legs Due to Venous Reflux
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1138.6
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency

ARMS (1):
- BNS003 (Experimental)
  Interventions: Drug: BNS003

INTERVENTIONS:
Drug: BNS003

SUMMARY:
To investigate the efficacy and safety of BNS003 on subjective symptoms such as sensation of heaviness/tiredness(dullness), tension, tingling, pain, fever or itching associated with swelling of calf and ankle due to disorder of leg venous reflux.

ELIGIBILITY:
Inclusion Criteria:

* Manifestation of swelling falling into Class 1 according to Porter's classification
* With more than 2 symptoms of "sensation of heaviness/tiredness (dullness)," "tension," "tingling," "pain," "fever" or "itching" and a total score of >=3 for severity by symptoms
* Persons aged 20 years or older at the time of obtaining their informed consent and available for hospital visits. Both genders are acceptable
* Persons who have consented to participating in the study in written form with good understanding of the objective of the study, the methods, and notices for the study period

Exclusion Criteria:

* Persons with edema not due to venous diseases of the legs (e.g., lymphedema, latent cardiac or renal insufficiency, etc.)
* Persons with peripheral arterial diseases
* Persons with acute phlebitis, venous ulcer, congenital vascular anomaly, or Behcet's Syndrome
* Persons with "moderate" or "severe" renal, hepatic, cardiac or haematological disorder, or with a history of such disorder (Grade 3 or 4 in Common Toxicity Criteria (CTC))
* Persons with diabetes mellitus (excluding those curable with dietary therapy), neuropathy, hyper-or hypocalcemia, or malignant tumors
* Persons with drug or alcohol abuse
* Persons with immobility
* Persons with pulmonary embolism
* Persons with hypersensitivity to drugs (particularly to the ingredients contained in the investigational drug)
* Persons with clinical indication of requiring venous treatment such as physical application (use of elastic bandage and compression stockings) and phlebectomy (vein stripping surgery to remove vein affected with varicosis and valve insufficiency)
* Persons who received venous sclerosing therapy within the last 4 weeks before starting this study
* Persons who constantly use theophylline preparations, diuretics, cardiac glycosides
* Persons who had changed to or initiated post-menopausal hormone replacement therapy within the last 2 months before starting this study
* Persons unable to suspend the frequent use and exceeded dosage/administration of laxatives (more than 6 times) during the study period
* Persons planned to undergo a surgery requiring systemic anesthesia during the study period
* Women in pregnancy or nursing, or those who wish for a pregnancy during the study period
* Persons who participated in another study within the last 3 months before starting this study, or who plan to participate in another study during the study period
* Persons who were considered to be ineligible to be a subject for the trial by the investigator or sub-investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2004-07; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Global improvement on a five point scale | week 12
  The degree of improvement was evaluated according to change of severity of each symptom at the time of enrollment (baseline) and in Week 12 after initiation of dosing (or at discontinuation)
Number of patients with adverse drug reactions | up to week 12

SECONDARY OUTCOMES:
Improvement per symptom on a five point scale | 12 weeks
Change in circumference measurements of calf in centimetres | baseline, 12 weeks
Change in circumference measurements of ankle in centimetres | baseline, 12 weeks
Subject's impression on improvement on a five point scale | baseline, 12 weeks
Number of patients with of adverse events | up to 12 weeks